CLINICAL TRIAL: NCT03602001
Title: Attentive Eating for Weight Loss: Proof of Concept Non-blinded Randomised Control Trial
Brief Title: Attentive Eating for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: University of Birmingham (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principle Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1905; ES/N00034X/1 (Other Grant/Funding Number: ESRC)
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Overweight and Obesity
Keywords: attentive eating; e-health; weight loss; food intake
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- attentive eating smartphone app group (Experimental): Participant's received the intervention 'Attentive eating smartphone application'. This is a smartphone application that encourages a more attentive eating style. Participants also received the 'Standard dietary advice and text tips' intervention. This consists of a standard dietary advice booklet, and weekly dietary advice tips by text message.
  Interventions: Behavioral: Attentive eating smartphone application.; Behavioral: Standard dietary advice and text tips.
- control group (Active Comparator): Participants received the 'Standard dietary advice and text tips' intervention. This consists of a standard dietary advice booklet, and weekly dietary advice tips by text message.
  Interventions: Behavioral: Standard dietary advice and text tips.

INTERVENTIONS:
Behavioral: Attentive eating smartphone application. — A smartphone application that encourages a more attentive eating style.
  Arms: attentive eating smartphone app group
Behavioral: Standard dietary advice and text tips. — Standard dietary advice for weight loss booklet and weekly text tips containing dietary advice.

SUMMARY:
This trial examined whether a smartphone application designed to encourage a more attentive eating style could help people to lose weight, compared to a control group.

DETAILED DESCRIPTION:
There is evidence that enhancing memory for recent eating and focusing attention on food being consumed influences later energy intake. Studies have shown that attending to food being eaten can reduce food intake. This has since been implemented into a smartphone based 'attentive eating' application. In a feasibility trial of this mobile phone application, adults with overweight or obesity were encouraged to eat attentively by photographing their meals and making satiety ratings after they had eaten. Participants were also required to review what else they had eaten that day before entering their next meal, with an overall aim of encouraging a more attentive eating style. Adherence data and qualitative interviews suggested that the mobile phone app was generally acceptable to participants and easy to use. Participants reported that they felt the application increased their awareness of what they had been eating. There was also an average weight loss of 1.5kg across the 4 week period that participants used the application for. Given that the previous feasibility trial included no control condition, the aim of the current trial was to examine initial proof of concept for effectiveness of an attentive eating smartphone weight loss application.

In the current study the investigators hypothesised that participants randomised to the attentive eating smartphone based condition (experimental condition) would lose significantly more weight than participants randomised to the control condition.

The study is a single centre, parallel, two arm, individually randomised 8 week controlled trial in adults with overweight and obesity in the Merseyside area of England.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25.0 kg/m2
* Self-report would like to lose weight by changing their dietary behaviour
* 18-65 years
* Fluent English
* Own an Android/Apple smartphone

Exclusion Criteria:

* History of eating disorders or food allergies
* Medication that affects appetite
* Pregnant
* Scheduled for weight loss survey during the trial
* Currently on a structured weight loss programme (e.g. Weight Watchers)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Weight at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Weight (kg) measured using Tanita Body composition scales. A lower body weight is considered a better outcome.
Self-reported energy intake at 4 weeks. | Measured at 4 weeks from the start of the trial.
  Energy intake (kcal) measured via 24HR recall. Lower energy intake is considered a better outcome.
Self-reported energy intake at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Energy intake (kcal) measured via 24HR recall. Lower energy intake is considered a better outcome.
Objective laboratory measured energy intake at 4 weeks. | Measured at 4 weeks from the start of the trial.
  Energy intake (kcal) measured with a bogus taste-test task. Lower energy intake is considered a better outcome.
Objective laboratory measured energy intake at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Energy intake (kcal) measured with a bogus taste-test task. Lower energy intake is considered a better outcome.

SECONDARY OUTCOMES:
Weight at 4 weeks. | Measured at 4 weeks from the start of the trial.
  Weight (kg) measured using Tanita Body composition scales. A lower body weight is considered a better outcome.
Body fat percentage at 4 weeks. | Measured at 4 weeks from the start of the trial.
  Body fat percentage measured using Tanita Body composition scales. A lower body fat percentage is considered a better outcome.
Body fat percentage at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Body fat percentage measured using Tanita Body composition scales. A lower body fat percentage is considered a better outcome.

OTHER OUTCOMES:
Ideal portion size at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Assessed using a computer-based visual portion size task, where participants will be asked to indicate their ideal serving size for 18 meals. In this task participants are shown portion size photographs of a meal on the screen, and are asked to use buttons on the keyboard to adjust the portion size. Based on their responses for the 18 meals, participants are assigned a value (in kcals) that represents the average energy content of their ideal portion size.
Uncontrolled eating measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  The Three Factor Eating Questionnaire-21 (Cappelleri et al., 2009) will be used to measure uncontrolled eating. The possible range of scores is 1-4 and higher scores indicate higher levels of uncontrolled eating. A lower score is considered a better outcome.
Cognitive restraint measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  The cognitive restraint sub-scale of the Three Factor Eating Questionnaire-21 will be used to measured cognitive restraint (Cappelleri et al., 2009). The possible range of scores is 1-4 and higher scores indicate higher levels of cognitive restraint. A lower score is considered a better outcome.
Emotional eating measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  The emotional eating sub scale of the Three Factor Eating Questionnaire-21 will be used to measured emotional eating (Cappelleri et al., 2009). The possible range of scores is 1-4 and higher scores indicate higher levels of emotional eating. A lower score is considered a better outcome.
Binge eating symptoms measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  The Binge Eating Scale will be used to measured binge eating symptoms (Gormally, Black, Daston, & Rardin, 1982). The possible range of scores is 0-46 and higher scores indicate a greater number of binge eating symptoms. A lower score is considered a better outcome.
Food cravings measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Food cravings will be measured using the Food Cravings Questionnaire (Nijs, Franken, & Muris, 2007). The possible range of scores is 21-126 and higher scores indicate a greater food cravings. A lower score is considered a better outcome.
Intuitive eating measured at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Intuitive eating will be measured using the reliance on hunger and satiety cues sub-scale of the Intuitive Eating Scale (IES-2; Tylka & Kroon Van Diest, 2013). The possible range of scores is 1-5, and higher scores indicate greater intuitive eating (and greater reliance on hunger and satiety signals). A higher score is considered a better outcome.
Intervention efficacy beliefs at baseline. | Measured at baseline.
  Participants beliefs about how confident they are that the intervention will help them to eat less and lose weight will be measured. The scale consists of 2 questions scored on 100-point visual analogue scales. If responses to both questions are strongly correlated (r ≥ 0.7), the average of the items will be computed to form a single composite measure. The possible score range is 0-100, with higher scores indicating higher beliefs that the intervention will help participants reduce food intake and aid weight loss.
Intervention efficacy beliefs at 8 weeks. | Measured at 8 weeks from the start of the trial.
  Participants beliefs about how confident they are that the intervention helped them to eat less and lose weight will be measured. The scale consists of 2 questions scored on 100-point visual analogue scales. If responses to both questions are strongly correlated (r ≥ 0.7), the average of the items will be computed to form a single composite measure. The possible score range is 0-100, with higher scores indicating higher beliefs that the intervention helped participants reduce their food intake and lose weight.
Smartphone application usage. | Data downloaded at 8 weeks from the start of the trial.
  At 8 week follow-up the researcher will download attentive eating application usage information. This will provide us with information about how often participants used the mobile phone application during the trial (e.g. number of times per day the application was accessed).
Semi-structured interviews at 8 weeks. | Conducted at 8 weeks from the start of the trial.
  Semi-structured interviews will be conducted with participants in the experimental group during the 8 week follow-up visit, in order to understand participants' experiences of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and statistical analysis plan were pre-registered prior to starting recruitment. IPD will be made available shortly prior to publication.
Access Criteria: The study protocol and statistical analysis plan were pre-registered prior to starting recruitment on the Open Science Framework, these can be accessed via this link. Datafile(s), including IPD, will be made publicly available here also. Link: https://osf.io/btzhw/
URL: https://osf.io/btzhw/

REFERENCES:
- [Background] Cappelleri JC, Bushmakin AG, Gerber RA, Leidy NK, Sexton CC, Lowe MR, Karlsson J. Psychometric analysis of the Three-Factor Eating Questionnaire-R21: results from a large diverse sample of obese and non-obese participants. Int J Obes (Lond). 2009 Jun;33(6):611-20. doi: 10.1038/ijo.2009.74. Epub 2009 Apr 28. PMID 19399021
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Nijs IM, Franken IH, Muris P. The modified Trait and State Food-Cravings Questionnaires: development and validation of a general index of food craving. Appetite. 2007 Jul;49(1):38-46. doi: 10.1016/j.appet.2006.11.001. Epub 2006 Dec 21. PMID 17187897
- [Background] Tylka TL, Kroon Van Diest AM. The Intuitive Eating Scale-2: item refinement and psychometric evaluation with college women and men. J Couns Psychol. 2013 Jan;60(1):137-53. doi: 10.1037/a0030893. PMID 23356469
- [Derived] Whitelock V, Kersbergen I, Higgs S, Aveyard P, Halford JC, Robinson E. User Experiences of a Smartphone-Based Attentive Eating App and Their Association With Diet and Weight Loss Outcomes: Thematic and Exploratory Analyses From a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Oct 2;8(10):e16780. doi: 10.2196/16780. PMID 33006564
- [Derived] Whitelock V, Kersbergen I, Higgs S, Aveyard P, Halford JCG, Robinson E. A smartphone based attentive eating intervention for energy intake and weight loss: results from a randomised controlled trial. BMC Public Health. 2019 May 21;19(1):611. doi: 10.1186/s12889-019-6923-x. PMID 31113400
- Available data/document: Study Protocol — https://osf.io/btzhw/ — The study protocol was pre-registered prior to starting recruitment on the Open Science Framework and is available via this link. IPD underlying publications will also be available here.